CLINICAL TRIAL: NCT03899454
Title: Randomized Clinical Trial of the Effect of G. Mangostana L Rind and Solanum Lycopersicum Fructus Extract to Prevent Exercise-induced Oxidative Stress
Brief Title: Garcinia Mangostana L Rind and Solanum Lycopersicum Fructus Trial to Prevent Exercise-induced Oxidative Stress
Acronym: GMR-RCT-EOS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitas Negeri Semarang (Other)
Collaborators: Ministry of Research, Technology and Higher Education, Republic of Indonesia (Unknown)
Responsible Party: Principal Investigator, Mahalul Azam, Principle Investigator, Universitas Negeri Semarang
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCT 201901
Record Dates: First submitted 2019-03-28; First posted 2019-04-02 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Exertion; Excess; Oxidative Stress
Keywords: exercise-induced oxidative-stress; Garcinia mangostana L rind

STUDY DESIGN:
Intervention Model Description: two arm treatment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extract administration (Experimental): administration of a mixed extract of Garcinia mangostana 400mg and Solanum Lycopersicum Fructus 200mg (OKSI(R) POM TR 193324351)
  Interventions: Drug: Garcinia-mangostana-L-rind and Solanum-Lycopersicum-Fructus mixture-extract
- Control (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Control

INTERVENTIONS:
Drug: Garcinia-mangostana-L-rind and Solanum-Lycopersicum-Fructus mixture-extract — Administration of mixed extract of Garcinia mangostana 400mg and Solanum Lycopersicum Fructus 200mg (OKSI(R) POM TR 193324351)
  Other Names: Brand name: OKSI (Indonesian Food and Drug Administration POM registered number :TR 193324351)
  Arms: Extract administration
Drug: Placebo Control — Placebo Control
  Other Names: placebo
  Arms: Control

SUMMARY:
Treatments are an administration of a mixed extract of Garcinia mangostana 400mg and Solanum Lycopersicum Fructus 200mg (OKSI(R) POM TR 193324351) and placebo control.

DETAILED DESCRIPTION:
Double-blinded Randomized Clinical Trial

The population of study will involve sedentary men, the student in Universitas Negeri Semarang aged 18-25 years old, targetted populations are 30 subjects consist of 15 treatment group and the rest 15 placebo-control group. Voluntary sampling will be conducted. Information to the candidates delivered directly, leaflets, and social media broadcasting.

Two arm treatment to be given is an administration of a mixture extract of Garcinia mangostana 400mg and Solanum Lycopersicum Fructus 200mg (OKSI(R) POM TR 193324351) and placebo control.

The administration of extract treatment and placebo will be given for four weeks.

The primary effect that will be observed is the changes in malondialdehyde (MDA) and high-sensitivity Cardiac-Troponin I (hs-cTnI) level after an ergo-cycle exercise test.

The secondary effect of the treatment that will be observed is the baseline and post-treatment parameters of MDA levels.

ELIGIBILITY:
Inclusion Criteria:

* sedentary lifestyle
* apparently healthy person
* willing to use the smart-phone application for diet and physical activity monitoring

Exclusion Criteria:

* pathological appearance in ECG

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07-15 (Estimated); Primary Completion 2020-09-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Change ergo-cycle exercise test response to MDA level after 4 weeks treatment | 4 weeks
  measuring exercise-induced oxidative stress, based on pre-and post-exercise MDA levels
Change ergo-cycle exercise test response to hs-cTnI level after 4 weeks treatment | 4 weeks
  measuring exercise-induced oxidative stress, based on pre-and post-exercise hs-cTnI levels

SECONDARY OUTCOMES:
Change from baseline MDA levels after 4 weeks treatment | 4 weeks
  measuring MDA levels baseline and post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mahalul Azam, Principal Investigator — Universitas Negeri Semarang
Locations (1):
- Universitas Negeri Semarang, Semarang, Central Java, Indonesia

REFERENCES:
- [Background] Knez WL, Jenkins DG, Coombes JS. Oxidative stress in half and full Ironman triathletes. Med Sci Sports Exerc. 2007 Feb;39(2):283-8. doi: 10.1249/01.mss.0000246999.09718.0c. PMID 17277592
- [Background] Thompson PD, Stern MP, Williams P, Duncan K, Haskell WL, Wood PD. Death during jogging or running. A study of 18 cases. JAMA. 1979 Sep 21;242(12):1265-7. PMID 480538
- [Background] Eijsvogels T, George K, Shave R, Gaze D, Levine BD, Hopman MT, Thijssen DH. Effect of prolonged walking on cardiac troponin levels. Am J Cardiol. 2010 Jan 15;105(2):267-72. doi: 10.1016/j.amjcard.2009.08.679. PMID 20102930
- [Background] Tong TK, Kong Z, Lin H, He Y, Lippi G, Shi Q, Zhang H, Nie J. Effects of 12-Week Endurance Training at Natural Low Altitude on the Blood Redox Homeostasis of Professional Adolescent Athletes: A Quasi-Experimental Field Trial. Oxid Med Cell Longev. 2016;2016:4848015. doi: 10.1155/2016/4848015. Epub 2015 Dec 10. PMID 26783415
- [Background] Tjahjani S, Widowati W, Khiong K, Suhendra A, Tjokropranoto R. Antioxidant Properties of Garcinia Mangostana L (Mangosteen) Rind. Procedia Chem. 2014
- [Background] Sutono, T. Efficacy of Garcinia mangostana L. (mangosteen rind extract) to reduce acne severity. Med J Indones. Vol. 22, No. 3, August 2013
- [Background] Meechai I, Phupong W, Chunglok W, Meepowpan P. Dihydroosajaxanthone: A New Natural Xanthone from the Branches of Garcinia Schomburgkiana Pierre. Iran J Pharm Res. 2018 Fall;17(4):1347-1352. PMID 30568693
- [Background] Ali Hassan SH, Fry JR, Abu Bakar MF. Phytochemicals content, antioxidant activity and acetylcholinesterase inhibition properties of indigenous Garcinia parvifolia fruit. Biomed Res Int. 2013;2013:138950. doi: 10.1155/2013/138950. Epub 2013 Oct 31. PMID 24288662